CLINICAL TRIAL: NCT03251833
Title: The Impact of Obesity on Maternal and Perinatal Outcomes; Analytic Cross Sectional Study
Brief Title: The Impact of Obesity on Maternal and Perinatal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: OMP
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese: Body mass index >30 Kilogram/m2
- non-obese: Body mass index <30 Kilogram/m2

SUMMARY:
Body Mass Index is an index that is commonly used to classify underweight, overweight and obesity in adults. It is defined as the weight in kilograms divided by the square of the height in meters.The growing epidemic of obesity in our society has become a major public health issue where the proportion of overweight and obese among women aged 15-59 have increased from 68 percent in 2008 to 76 percent in 2015

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* single fetus
* gestational age >28weeks

Exclusion Criteria:

* patient refusal
* multifetal pregnancy
* Medical illness prior to pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women admitted to the emergency unit of Obstetrics and Gynaecology Department, Woman's Health Hospital
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-03-04 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of preeclampsia in both groups | 24 hours
  The number of women who develop hypertension with proteinuria in pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No